CLINICAL TRIAL: NCT04213274
Title: A Randomized, Double-Blind, Placebo-Controlled, Multicenter, Phase 2 Study of the Efficacy and Safety of RPH-104 in Adult Subjects With Schnitzler Syndrome
Brief Title: Study of the Efficacy and Safety of RPH-104 in Adult Subjects With Schnitzler Syndrome
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: due to the decision of company Top management
Sponsor: R-Pharm Overseas, Inc. (Industry)
Collaborators: Worldwide Clinical Trials (Other)
Responsible Party: Sponsor
Organization: R-Pharm (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CL04018066
Record Dates: First submitted 2019-10-22; First posted 2019-12-30 (Actual); Last update posted 2024-11-15 (Actual); Status verified 2024-11

CONDITIONS: Schnitzler Syndrome; Urticarial Vasculitis With Monoclonal Immunoglobulin M Component, Schnitzler (Disorder)
Keywords: neutrophilic urticarial dermatosis; autoinflammatory syndrome; monoclonal gammopathy; neutrophilic dermatosis; interleukin-1; Schnitzler syndrome
MeSH Terms: conditions — Schnitzler Syndrome; Paraproteinemias

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Placebo - placebo (Placebo Comparator): Subject randomized to receive subcutaneous single injection of placebo on Day 0,and then, on Day 14 - second dose of randomized treatment + based on the positive response to treatment (SDAS = 0) one more dose of placebo
  Interventions: Drug: Placebo
- Placebo - 80 mg RPH-104 (Other): Subject randomized to receive subcutaneous single injection of placebo on Day 0,and then, on Day 14 - second dose of randomized treatment + based on the lack of response (no change in SDAS) or partial response to treatment (SDAS ≥ 1, and activity reduction by 1 or more points of SDAS compared to baseline) subcutaneous single injection of 80 mg RPH-104
  Interventions: Biological: 80 mg RPH-104; Drug: Placebo
- 80 mg RPH-104 - 80 mg RPH-104 (Experimental): Subject randomized to receive subcutaneous single injection of 80 mg RPH-104 on Day 0,and then, on Day 14 - second dose of randomized treatment + based on the positive response to the treatment (SDAS = 0) one subcutaneous injection of placebo
  Interventions: Biological: 80 mg RPH-104; Drug: Placebo
- 80 mg RPH-104 - 160 mg RPH-104 (Experimental): Subject randomized to receive subcutaneous single injection of 80 mg RPH-104 on Day 0,and then, on Day 14 - second dose of randomized treatment + based on the lack of response (no change in SDAS) or partial response to treatment (SDAS ≥ 1, and activity reduction by 1 or more points of SDAS compared to baseline) one more subcutaneous injection of 80 mg RPH-104
  Interventions: Biological: 80 mg RPH-104

INTERVENTIONS:
Biological: 80 mg RPH-104 — solution for subcutaneous administration 40 mg/mL, 2 mL in the 4-mL glass vial
  Arms: 80 mg RPH-104 - 160 mg RPH-104; 80 mg RPH-104 - 80 mg RPH-104; Placebo - 80 mg RPH-104
Drug: Placebo — Normal Saline (0.9% Sodium Chloride solution for Injection), 2 mL in the 4 mL-glass vial
  Arms: 80 mg RPH-104 - 80 mg RPH-104; Placebo - 80 mg RPH-104; Placebo - placebo

SUMMARY:
The primary goal of the study is to assess the efficacy and safety of RPH-104 in subjects with Schnitzler Syndrome using Schnitzler Disease Activity Score (SDAS), which includes the Physician's Global Assessment (PGA) and the local laboratory C-reactive protein (CRP) result

DETAILED DESCRIPTION:
The study will include a screening period (up to 28 days), a double blind, placebo controlled treatment period (14 days), followed by an 8 week safety follow up period after the second dose of study drug.

Subjects with an established diagnosis of Schnitzler Syndrome (SchS) will participate in a Screening period of up to 28 days after signing an informed consent form (ICF). Subjects will be advised to schedule the Day 0 visit with the study staff as soon as the symptoms of SchS flare occur during the Screening period.

If the subject does not meet the inclusion/exclusion criteria at the site visit during the screening period, other screening visits are allowed within this period until the subject meets the study criteria.

A total of 14 subjects will be randomly assigned to 1 of 2 treatment groups (in a 1:1 ratio) to receive a double blind, single subcutaneous (SC) injection of study drug (80 mg RPH-104 or matching placebo) on Day 0. On Day 14, subjects will receive a second dose of randomized treatment as well as an additional dose of 80 mg RPH-104 or placebo based on response to treatment, such that responders (SDAS = 0) will receive a dose of placebo, and non responders defined as no response (no change in SDAS) or partial responders (SDAS ≥ 1, and activity reduction by 1 or more points of SDAS compared to baseline) will receive an 80 mg RPH 104 dose. (Schnitzler Disease Activity Score includes the PGA score and C-reactive protein (CRP) result: If the PGA and CRP grades are not of the same severity, the higher severity level of either PGA or CRP will be used to determine the SDAS)

The study will be stopped after Data and Safety Monitoring Board (DSMB) review if:

1. Death is reported in 2 subjects assigned to the RPH 104 treatment arm or after receiving RPH 104 on Day 14 (i.e., non responder to the Day 0 study drug dose).
2. Two subjects assigned to the RPH 104 treatment arm or after receiving RPH 104 on Day 14 (ie, non responder to the Day 0 study drug dose) report liver function test abnormalities which meet Hy's Law criteria (ie, increased ALT and/or AST 3 fold or greater from upper limit of normal (ULN) combined with jaundice or weakness or hypochondrial pain/severity or increased Total Bilirubin (TBil) level 2 fold or greater from ULN, [not explained by any other causative factors like virus]).

The severity of SchS symptoms will be assessed daily from Day 0 through Day 28 using the PR SchS Scale, at clinic visits on Day 0, Day 14, and Day 28 using the Patient Global Impression of Severity (PGIS), at clinic visits on Day 14 and Day 28 using the Patient Global Impression of Change (PGIC), and at each clinic visit using the PGA, CRP, SAA, and SDAS. Subjects will be followed through Day 70 for safety (A Data Safety Monitoring Board (DSMB) will periodically review and evaluate the accumulated study data for subject safety).

ELIGIBILITY:
Inclusion Criteria:

* 1. Able to read, understand and willing to sign the ICF and abide with study procedures. The ICF must be signed and dated prior to performing any Screening assessment.
* 2. Confirmed diagnosis of SchS based on diagnostic criteria adapted by Lipsker as an urticarial skin rash (chronic), monoclonal IgM component (ie, IgM < 10 g/L), or IgG (variant type), and at least of 2 of the following:

  * Fever (intermittent)
  * Arthralgia or arthritis
  * Bone pain
  * Lymphadenopathy
  * Hepato and/or splenomegaly
  * Elevated erythrocyte sedimentation rate (ESR) and/or leukocytosis
  * Bone abnormalities (on radiological or histological investigation)
* 3. Subjects with symptomatic SchS (as defined by SDAS with a score of 2 or more with a CRP [local laboratory] levels > 10 mg/L) on the day of randomization.
* 4. Willing, committed, and able to return for all clinic visits and complete all study related procedures, including willingness to have SC injections administered by a qualified person.
* 5. Males, female partners of sexually active male subjects, and women of childbearing potential (WOCBP) (defined as all female subjects with physiological potential to conceive) must agree to use highly effective contraceptive methods throughout the study starting from Screening (signing informed consent) through at least 8 weeks after the final dose of study drug.

Highly effective contraceptive method is defined as follows:

1. Complete abstinence: if it corresponds to the preferred and conventional lifestyle of the female subject. Periodic abstinence (eg, calendar, ovulation, symptothermal, postovulation method) and interrupted coitus are not considered acceptable contraceptive methods.
2. Sterilization: surgical bilateral ovariectomy (with/without hysterectomy) or tubal ligation at least 6 weeks prior to the study therapy initiation. In case of ovariectomy only the female reproductive status should be verified by further hormonal test.
3. Sterilization of male partner with documented absence of sperm in ejaculate post vasectomy for at least 6 months (vasectomized male partner should be the only partner of the participating female subject).
4. Combination of 2 of the following methods (i + ii, i + iii, or ii + iii):

i. Oral, injectable, or implanted hormonal contraceptives; in case of oral contraceptives the female subjects should administer the same product for at least 3 months prior to the study therapy.

ii. Intrauterine device or contraceptive system.

iii. Barrier methods: condom or occlusive cap (diaphragm or cervical cap/vaginal fornix cap) with spermicidal foam/gel/film/cream/vaginal suppository.

* 6. WOCBP must have negative pregnancy tests at Screening (serum chorionic gonadotropin test), and all subsequent visits (urine).

Exclusion Criteria:

* 1. Hypersensitivity to the study drug (RPH 104) and/or its components/excipients and/or the products of the same chemical class.
* 2. Concurrent/on going treatment with anakinra (Kineret) or recent treatment within 5 days prior to Day 0.
* 3. Concurrent/on going treatment with other biologics or recent treatment within 4 weeks or 5 × t½ prior to Day 0, whichever is longer.
* 4. Concurrent/on going treatment with immunosuppressive agents (eg, cyclosporine, methotrexate, dapsone, colchicine, or others) within 4 weeks or 5 × t½ prior to Day 0, whichever is longer.
* 5. Concurrent/on going treatment with high doses of systemic steroids (> 0.2 mg/kg/day prednisolone equivalent). Intra articular, peri articular, intravenous, or intramuscular corticosteroid injections within 4 weeks prior to the Day 0 visit.
* 6. Administration of live (attenuated) vaccine within 3 months prior to Day 0 and necessity of live vaccine administration for 3 months after Day 70.
* 7.

  1. History of active tuberculosis (TB), evidence of active or latent M. tuberculosis infection as defined by local guidelines/local medical practice at Screening.
  2. Positive QuantiFERON Gold Plus (TB) test at Screening.
  3. Chest X ray findings confirming pulmonary TB at Screening.
* 8. Active bacterial, fungal, or viral infection(s) within 4 weeks prior to Day 0.
* 9. A history of persistent chronic bacterial, fungal, or viral infection(s) requiring treatment with parenteral antibiotics, parenteral antivirals, or parenteral antifungals within 4 weeks prior to Day 0.
* 10. Opportunistic infections and/or Kaposi's sarcoma at the time of Screening.
* 11. Any other relevant concomitant diseases (infectious, cardiovascular, nervous, endocrine, urinary, gastrointestinal, hepatic disorders, coagulation disorders, and other autoimmune/autoinflammatory diseases, etc) or conditions which, according to the investigator's judgment, may affect the subject's participation or well being in the study and/or distort assessment of the study results.
* 12. History of malignancies within 5 years prior to screening other than successfully treated non metastatic, basal, or squamous cell carcinoma of the skin and/or in situ cancer.
* 13. Evidence of lymphoproliferative diseases (except SchS associated monoclonal gammopathy).
* 14. Presence of any of the following laboratory abnormalities at screening visit: white blood cell count (WBC) < 3000/µL; platelet count < 75,000/µL; alanine aminotransferase (ALT) or aspartate aminotransferase (AST) > 3.0 × upper limit of normal (ULN), TBil > 2 × ULN unless due to Gilbert's syndrome.
* 15. Severe renal failure: Cockcroft Gault creatinine clearance < 30 mL/min.
* 16. Women who are either pregnant or lactating.
* 17. Subjects for whom there is concern about compliance with the protocol procedures.
* 18. Psychiatric disorders which, according to the investigator's judgment, may affect the subject participation in the study and his/her ability to follow the protocol procedures.
* 19. History of organ transplantation or transplantation is anticipated during the study.
* 20. Concomitant participation in other clinical studies at the start of Screening or administration of any unauthorized (investigational) products less than 4 weeks or 5 × t½ periods (whichever is longer) before Day 0 (treatment initiation).

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-05 (Estimated); Primary Completion 2023-08 (Estimated); Study Completion 2024-01 (Estimated)

PRIMARY OUTCOMES:
Proportion of subjects with complete response (Schnitzler Disease Activity Score (SDAS = 0)) to therapy on Day 14 in the RPH-104 group as compared to the placebo group | Day 14
  • Proportion of subjects with complete response (SDAS = 0) to therapy on Day 14 in the RPH 104 treated group as compared to the placebo group based on SDAS using the PGA and the local laboratory CRP result

SECONDARY OUTCOMES:
Change from baseline to Day 14 in subject-reported symptom severity of SchS: Patient-reported Severity of Schnitzler Syndrome Scale (PR-SchS Scale) | Baseline and Day 14
  Change from baseline to Day 14 in subject-reported symptom severity of SchS using the Patient-reported Severity of Schnitzler Syndrome Scale (PR-SchS Scale). The PR-SchS Scale includes 5 features that are the most common and important SchS symptoms. These include rash, fever, tiredness, joint pain, and bone/muscle pain.
Proportion of subjects with normalized serum amyloid A (SAA) and C-reactive protein (CRP) at Days 14 and 28 | Day 14 and Day 28
  Proportion of subjects with normalized SAA (< 10 mg/L) and CRP (≤ 10 mg/L) at Days 14 and 28
Change from baseline to Day 14 and Day 28 in CRP and SAA | Baseline, Day 28 and Day 14
  Change from baseline to Day 14 and Day 28 in C-reactive protein and serum amyloid A
Proportion of subjects with complete response (SDAS = 0) to therapy on Day 28 by treatment sequence based on SDAS using the Physician's Global Assessment (PGA) and the CRP result | Baseline and Day 28
  Proportion of subjects with complete response (SDAS = 0) to therapy on Day 28 by treatment sequence (placebo - placebo, placebo - 80 mg RPH 104, 80 mg RPH 104 80 mg RPH 104, and 80 mg RPH 104 - 160 mg RPH 104) based on SDAS using the PGA and the CRP result.
Proportion of subjects with partial response by treatment sequence on Days 14 and 28 | Baseline, Day 14 and Day 28
  Proportion of subjects with partial response (SDAS ≥ 1, and activity reduction by 1 or more points of SDAS compared to baseline) by treatment sequence (placebo - placebo, placebo 80 mg RPH 104, 80 mg RPH 104 80 mg RPH 104, and 80 mg RPH 104 160 mg RPH 104) on Days 14 and 28

OTHER OUTCOMES:
Change from baseline to Day 28 in subject reported symptom severity of SchS using the PR SchS Scale | Baseline, Day 14 and Day 28
  Change from baseline to Day 28 in subject reported symptom severity of SchS using the PR SchS Scale
Change from baseline to Day 14 and Day 28 in the Short Form-36 Version 2 Health Survey® | Baseline, Day 14 and Day 28
  Change from baseline to Day 14 and Day 28 in the Short Form-36 Version 2 Health Survey® (SF 36v2 scale scores).It should be completed by the subject to assess of their quality of life over the preceding week.The SF 36v2 is a 36 item, patient reported survey of patient health. It consists of 8 health domains, including: Vitality,Physical functioning,Bodily pain, General health perceptions, Physical role functioning, Emotional role functioning, Social role functioning, Mental health.The SF 36v2 also produces 2 summary scores: the physical component summary (PCS) and mental component summary (MCS) scores
Change from baseline to Day 14 and Day 28 in PGA total score | Baseline, Day 14 and Day 28
  Change from baseline to Day 14 and Day 28 in PGA (Physician's Global Assessment) total score. 5 key symptoms of SchS (urticarial rash, fatigue, fever, myalgia, and arthralgia/bone pain) will be evaluated with a PGA score. Each symptom to be graded on a 4-point Likert scale where 0 = no, 1 = mild, 2 = moderate, and 3 = severe disease activity. The total PGA score to be ranged between 0 and 15.
Change from baseline to Day 14 and Day 28 in PGIS scores | Baseline, Day 14 and Day 28
  Change from baseline to Day 14 and Day 28 in PGIS scores (Patient Global Impression of Severity score: The PGIS asks subjects to describe the severity of their symptoms right now.Subjects are asked: "Please choose the response below that best describes the severity of your Schnitzler Syndrome symptoms today". Subjects rate their symptoms on a 5-point scale as "None", "Mild", "Moderate", "Severe", or "Very Severe")
Proportion of subjects who are "Much Better" or "A Little Better" in PGIC scores at Day 14 and Day 28 | Day 14 and Day 28
  Proportion of subjects who are "Much Better" or "A Little Better" in PGIC scores at Day 14 and Day 28. (PGIC is a 5-point scale, where the subjects should rate the overall change in their symptoms by comparing the severity of their symptoms right now with the severity of their symptoms before they began study treatment. Subjects are asked: "Please choose the response below that best describes the overall change in your Schnitzler Syndrome symptoms since you started taking the study medication". Subjects report their change in symptoms as "Much better","A Little Better", "No Change", "A Little Worse", or "Much worse")
Change from baseline to Day 14 and Day 28 in IgG levels | Baseline, Day 14 and Day 28
  Change from baseline to Day 14 and Day 28 in immunoglobulin G (IgG) levels
Change from baseline to Day 14 and Day 28 in IgM levels | Baseline, Day 14 and Day 28
  Change from baseline to Day 14 and Day 28 in immunoglobulin M (IgM) levels
Change from baseline to Day 14 and Day 28 in IgA levels | Baseline, Day 14 and Day 28
  Change from baseline to Day 14 and Day 28 in Immunoglobulin A (IgA) levels
Change from baseline to Day 14 and Day 28 in Kappa protein levels | Baseline, Day 14 and Day 28
  Change from baseline to Day 14 and Day 28 in Kappa protein levels
Change from baseline to Day 14 and Day 28 in Lambda protein levels | Baseline, Day 14 and Day 28
  Change from baseline to Day 14 and Day 28 in Lambda protein levels
Change from baseline to Day 14 and Day 28 in Paraprotein levels | Baseline, Day 14 and Day 28
  Change from baseline to Day 14 and Day 28 in Paraprotein levels
Change from baseline to Day 14 and Day 28 in Binding and neutralizing antidrug antibodies levels | Baseline, Day 14 and Day 28
  Change from baseline to Day 14 and Day 28 in Binding and neutralizing antidrug antibodies levels
Estimated half-life (t½) of RPH 104 | Baseline, Day 14, Day 28, Day 42, Day 70
  Estimated t½ of RPH 104
Change from baseline to Day 14 and Day 28 in IL-1β, IL-1α, IL-1RA, and IL-6 levels | Baseline, Day 14 and Day 28
  Change from baseline to Day 14 and Day 28 in IL-1β, IL-1α, IL-1 receptor antagonist (IL-1RA), and IL-6 levels
Viral testing at Screening | Screening
  Hepatitis B virus (HBV), hepatitis C virus (HCV), and human immunodeficiency virus (HIV) presence will be assessed
QuantiFERON Gold Plus (TB) test at Screening | Screening
  evidence of no active or latent M. tuberculosis infection as defined by local guidelines/local medical practice
Pregnancy test for all WOCBP (women of childbearing potential) | Screening, Baseline, Day 14, Day 28, Day 42, and Day 70
  serum chorionic gonadotropin test will be performed at screening and urine tests will be done at Baseline, Day 14, Day 28, Day 42, and Day 70
Change in CRP (C-reactive protein) test results from screening to Day 28 | Screening, Baseline, Day 14, Day 28
  CRP will be performed at both a local laboratory and the central laboratory. The local laboratory CRP test is to be processed on the same day the clinical assessments occur. Dosing cannot occur until these results are available on Day 0 and Day 14 to ensure eligibility and response to treatment.
Change in monoclonal proteins levels from baseline to Day 70 | Baseline, Day 14, Day 28, Day 42, and Day 70
  IgG, IgM, IgA, kappa, lambda, and paraprotein levels will be assessed
Change in SAA (serum amyloid A) test results from Screening to Day 70 | Screening, Baseline, Day 14, Day 28, Day 42, and Day 70
  Serum levels of SAA have been found to be elevated in SchS, and systemic AA amyloidosis as a consequence of chronic inflammation has been reported in SchS.The SAA analysis will be performed at the central laboratory

CONTACTS AND LOCATIONS:
Overall Officials: Yan Lavrovsky, Study Director — R-Pharm Overseas, Inc.
Locations (4):
- United States (4):
  - National Jewish Health, Denver, Colorado
  - Mayo Clinic, Rochester, Minnesota
  - Oregon Health & Science University, Portland, Oregon
  - Penn State Health Hersey Medical Center, Hershey, Pennsylvania